CLINICAL TRIAL: NCT06436183
Title: A Phase 2a, Multicenter, Randomized, Double-blind, 16-week Placebo-controlled Study With an Open Label Extension to Evaluate the Efficacy and Safety of Camoteskimab in Adults With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of the Effects of Camoteskimab in Adults With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apollo Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP43CP03
Record Dates: First submitted 2024-04-09; First posted 2024-05-30 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Atopic Dermatitis; Atopic; Dermatitis; Dermatologic Disease; Eczema; Eczema Atopic Dermatitis; Eczema, Atopic
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Skin Diseases; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental): Camoteskimab
  Interventions: Drug: Camoteskimab
- Dose 2 (Experimental): Camoteskimab
  Interventions: Drug: Camoteskimab; Drug: Placebo
- Placebo (Placebo Comparator): Dummy version of the study drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Camoteskimab — Drug Product
  Other Names: APL-9109; AVTX-007; CERC-007; AEVI-007; MEDI2338
  Arms: Dose 1; Dose 2
Drug: Placebo — Inactive substance
  Arms: Dose 2; Placebo

SUMMARY:
This is a Phase 2a, multicenter, randomized, double-blind, placebo-controlled study with an open-label extension to evaluate the efficacy and safety of camoteskimab in adults with moderate to severe AD.

DETAILED DESCRIPTION:
This study contains two parts: Parts 1 and Part 2.

Part 1 (Blinded Period):

Eligible patients will be randomized in a 1:1:1 ratio to receive either camoteskimab dose 1, camoteskimab dose 2 or placebo.

Part 2 (Extension Period):

In part 2, all participants will receive camoteskimab.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18-75 years of age inclusive, at the time of signing the informed consent.
2. Chronic AD for at least 1 year.
3. Participants with moderate to severe AD defined by:

   1. Investigator global assessment (IGA) score of ≥ 3 (on a scale of 0 to 4, in which three is moderate and four is severe) at Baseline.
   2. AD involvement of ≥ 10% body surface area (BSA) at Baseline.
   3. EASI score of ≥ 12 at Baseline.
   4. Pruritus numerical rating scale (NRS) ≥ 4 at Baseline.
4. Participants who are candidates for systemic therapy, defined as inadequate response to treatment with topical medications, or for whom topical treatments are otherwise medically inadvisable.
5. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Female participants:
   * Sexually active females of childbearing potential must agree to use two forms of accepted methods of highly effective forms of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes:
   * IUD plus one barrier method.
   * Stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method.
   * 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or
   * A vasectomized partner*.

   Male participants:
   * Sexually active male participants and males and who are partners of females of childbearing potential agree to use two forms of contraception as above and to not donate sperm or try to conceive during the treatment period and for at least 3 months after the last dose of study drug.
6. Participant provides signed informed consent.

Exclusion Criteria:

1. Participant has history of use of more than two (2) prior systemic therapies for AD (e.g.

   biologics or JAKi) and who used any of these medications as follows:
   1. Dupilumab, tralokinumab, lebrikizumab within 8 weeks prior to Baseline.
   2. Systemic JAKi within 4 weeks prior to Baseline.
   3. TCS, TCI, topical phosphodiesterase-4 (PDE4) inhibitors, and topical JAKi within 7 days prior to enrollment (at Baseline) or more than five half-lives whichever is longer.
2. Participant has a current diagnosis of other active skin disease (e.g., psoriasis or lupus erythematosus) or skin infection (bacterial, fungal, or viral) that may affect the evaluation of AD or would interfere with the study assessments.
3. Participant has a severe comorbidity that may require systemic steroids therapy or other interventions or requires active frequent monitoring (e.g., unstable chronic asthma).
4. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically significant abnormalities in the 12- lead ECG as considered by the perfusion index that may interfere with the interpretation of QTc interval changes.
5. Participant has AD involving ocular symptoms, or blepharitis, conjunctivitis, or keratitis diagnosed within the last 60 days prior to the screening visit, requiring chronic ocular corticosteroid treatment.
6. Participant has severe or uncontrolled seasonal or allergic rhinitis, asthma or any other non-AD disease as judged by the Investigator. Participants with seasonal or allergic rhinitis, asthma or any other non-AD disease requiring use of intranasal or inhaled corticosteroid that is stable and well-controlled are not excluded.
7. Active human immunodeficiency virus (HIV): confirmed positive anti-HIV antibody (HIV Ab) test; Active hepatitis B virus (HBV): confirmed hepatitis B surface antigen (HBs Ag) positive (+) or hepatitis B core antibody (HBc Ab) positive (+); Active hepatitis C virus (HCV): Confirmed hepatitis C antibody positive (+); evidence of active or latent TB
8. Diagnosed with a malignancy within 5 years of enrollment (suspected malignancy should be ruled out by blood or tissue biopsy, as applicable) with the exception of

   * Completely resected basal call or squamous cell carcinoma of the skin.
   * Carcinoma in situ of the cervix.
9. Has had previous exposure to anti-IL-18 therapy.
10. Treatment with any investigational agent, or any investigational device or procedure, within 28 days (or 5 half- lives, whichever is greater) of screening.
11. Has any of the following laboratory findings

    1. Glomerular filtration rate (GFR) < 30 mL/min/1.73 m2.
    2. Hemoglobin ≤8 g/dL.
    3. Neutrophils ≤1,500/μL.
    4. Platelets ≤75,000/μL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in Eczema Area and Severity Index (EASI) between camoteskimab and placebo at Week 12 | 12 weeks
  An EASI score is a tool used to measure the extent (area) and severity of atopic eczema. The EASI utilizes area assessments that rate the four involved regions on a 0% to 100% scale for each region. The scores are added up for each of the four body regions (head, arms, trunk, and legs). For each of these components, the individual scores are added together to calculate the EASI score, which ranges from 0 to 72. The higher the EASI score, the more severe the AD.

SECONDARY OUTCOMES:
Percent change from baseline in EASI score at Week 12 | 12 Weeks
  To further assess the efficacy of camoteskimab in participants with AD via the Eczema Area and Severity Index (EASI) which measures the severity of clinical signs in atopic dermatitis (AD).
Change from baseline in EASI score at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via the Eczema Area and Severity Index (EASI) which measures the severity of clinical signs in atopic dermatitis (AD).
Proportion of participants achieving a 50, 75, 90 and 100% improvement from baseline in EASI (EASI-50, 75, 90 and 100) at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via the Eczema Area and Severity Index (EASI) which measures the severity of clinical signs in atopic dermatitis (AD).
Proportion of participants with an IGA 0/1 and a decrease in IGA of ≥ 2 points at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via Investigator's Global Assessment Scale (IGA), which provides a global clinical assessment of AD severity.
Change from baseline in peak pruritus score at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via the Pruritus Numerical Rating Scale, which assesses itch severity.
Proportion of participants with an improvement of ≥ 4 or more points in peak pruritus weekly score at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via the Pruritus Numerical Rating Scale, which assesses itch severity.
Change from baseline in POEM score at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via the Patient-Oriented Eczema Measure (POEM) which assesses disease systems.
Change from baseline in DLQI score at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via the Dermatology Life Quality Index (DLQI) which assesses quality of life.
Change from baseline in AD involvement by BSA at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via Body Surface Area (BSA) which assesses the percentage of the total skin affected by AD.
Change from baseline in SP-NRS at Week 12 | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via the Skin Pain Numerical Rating Scale (SP-NRS) which assesses skin pain.
Change from baseline in PROMIS-SRI-SF-8a score at Week 12 reported outcomes | 12 weeks
  To further assess the efficacy of camoteskimab in participants with AD via Patient Reported Outcomes Measurement Information System (PROMIS) which measures patient-reported health status for physical, mental, and social well-being.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (30):
  - Medical Dermatology Specialists, PC/US Dermatology Partners, Phoenix, Arizona
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology Research, Inc., Fountain Valley, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - University of California Los Angeles Dermatology, Los Angeles, California
  - Amicis Research Center (Northridge), Northridge, California
  - Cura Clinical Research, Oxnard, California
  - VASDHS - Veterans Affairs San Diego Medical Center, San Diego, California
  - Clinical Sciences Institute, Santa Monica, California
  - Renaissance Research and Medical Group, Cape Coral, Florida
  - D&H National Research Centers, Inc., Miami, Florida
  - Avita Clinical Research - Dermatology, Tampa, Florida
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Owensboro Dermatology Associates, Owensboro, Kentucky
  - Revival Research Institute, Troy, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Michigan Dermatology Institute, Waterford, Michigan
  - Advanced Dermatology and Skin Cancer Center - Saint Joseph, Saint Joseph, Missouri
  - Skin Specialists PC, Omaha, Nebraska
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - ObjectiveHealth-The Skin Surgery Center for Clinical Research, Winston-Salem, North Carolina
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Unity Clinical Research - Dermatology, Oklahoma City, Oklahoma
  - Paddington Testing Co. Inc, Philadelphia, Pennsylvania
  - Rodgers Dermatology, Frisco, Texas
  - Center for Clinical Studies, Houston, Texas
  - Clinical Trial Network, Houston, Texas
- Canada (5):
  - Youthful Image, Edmonton, Alberta
  - Rejuvenation Dermatology Clinic Edmonton South, Edmonton, Alberta
  - Kingsway Clinical Research, Etobicoke, Ontario
  - Clinique Medicale Saint-Louis, Québec, Quebec
  - Clinique Dermatologique de Sherbrooke, Sherbrooke, Quebec